CLINICAL TRIAL: NCT06272500
Title: Safety and Efficacy Study of Betaine Hydrochloride in Treating Hypergastrinemia in Patients With Autoimmune Gastritis.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jianning Yao (Other)
Responsible Party: Sponsor-Investigator, Jianning Yao, Deputy Chief Physician, The First Affiliated Hospital of Zhengzhou University
Organization: The First Affiliated Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-KY-0146-001
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Autoimmune Gastritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo group (Placebo Comparator): receives oral administration of placebo, with two capsules before each meal.
  Interventions: Other: oral administration of receives only oral administration of placebo
- Betaine HCl Group (Experimental): receives oral administration of Betaine hydrochloride（BHCL), with two capsules before each meal.
  Interventions: Dietary Supplement: oral administration of Betaine hydrochloride

INTERVENTIONS:
Other: oral administration of receives only oral administration of placebo — receives oral administration of placebo, with two capsules before each meal.
  Arms: placebo group
Dietary Supplement: oral administration of Betaine hydrochloride — receives oral administration of Betaine hydrochloride(BHCL), with two capsules before each meal.
  Arms: Betaine HCl Group

SUMMARY:
Autoimmune atrophic gastritis (AAG) is an organ-specific autoimmune disease that primarily affects the gastric body and fundus while sparing the antrum. Its characteristics include destruction of gastric wall cells, loss of intrinsic factors, and atrophy of the gastric mucosa. Endoscopic examination reveals features of reverse atrophy, with significant atrophy in the gastric body and fundus, appearing as a mosaic of red and white patches. Currently, AAG is believed to result from a pathological CD4+ T-cell-mediated autoimmune response against the gastric H+/K+-ATPase. CD4+ T lymphocytes target the parietal cells' H+/K+-ATPase, stimulating plasma cells to secrete autoantibodies, including parietal cell antibodies (PCA) and intrinsic factor antibodies (IFA). The former plays a key role in parietal cell destruction and glandular atrophy. AAG is considered a premalignant condition, with the potential development of gastric dysplasia, cancer, and type 1 gastric neuroendocrine tumours (type 1 g-NET).

Gastric neuroendocrine tumors (g-NETs), also known as gastric carcinoids, account for approximately 23% of gastrointestinal and pancreatic neuroendocrine tumors. Clinically, g-NETs are mainly classified into three types. Type III is typically sporadic tumors associated with normal gastrin levels and poor prognosis. Although type 1 g-NETs caused by AAG are usually well-differentiated, studies have reported that 8%-23% of type 1 g-NETs extending into the deep submucosal layer may metastasize to regional lymph nodes or even to the liver. Furthermore, 3% of patients may develop neuroendocrine carcinoma, highlighting the need for appropriate attention.

Due to the destruction of gastric glands (including parietal and chief cells) in AAG patients, there is a deficiency in intrinsic factor, gastric acid, and a decrease in pepsinogen I (PG-I) levels. Insufficient gastric acid secretion leads to a compensatory increase in gastrin secretion by G cells in the gastric antrum, which acts on receptors present in enterochromaffin-like cells (ECL) in the gastric body and fundus, promoting ECL cell proliferation. Prolonged stimulation by hypergastrinemia can result in the development of ECL cell tumors, namely type 1 g-NETs. Considering the close association between type 1 g-NETs and AAG, primarily related to hypergastrinemia resulting from reduced gastric acid secretion, it is hypothesized that supplementation with gastric acid could provide negative feedback regulation of gastrin, reducing the risk of type 1 g-NET development in AAG patients. This study aims to investigate the impact of Betaine hydrochloride(BHCL) on gastrin levels in AAG patients, thus exploring a simple and cost-effective method to reduce the risk of type 1 g-NETs in AAG patients.

DETAILED DESCRIPTION:
Autoimmune atrophic gastritis (AAG) is an organ-specific autoimmune disease that primarily affects the gastric body and fundus while sparing the antrum. Its characteristics include destruction of gastric wall cells, loss of intrinsic factors, and atrophy of the gastric mucosa. Endoscopic examination reveals features of reverse atrophy, with significant atrophy in the gastric body and fundus, appearing as a mosaic of red and white patches, predominantly white, with flattened and partially disappearing folds and visible blood vessels. Currently, AAG is believed to result from a pathological CD4+ T-cell-mediated autoimmune response against the gastric H+/K+-ATPase. CD4+ T lymphocytes target the parietal cells' H+/K+-ATPase, stimulating plasma cells to secrete autoantibodies, including parietal cell antibodies (PCA) and intrinsic factor antibodies (IFA). The former plays a key role in parietal cell destruction and glandular atrophy, while the latter is the main mechanism underlying vitamin B12 deficiency and pernicious anaemia. AAG is considered a premalignant condition, with the potential development of gastric dysplasia, cancer, and type 1 gastric neuroendocrine tumours (type 1 g-NET).

Gastric neuroendocrine tumors (g-NETs), also known as gastric carcinoids, account for approximately 23% of gastrointestinal and pancreatic neuroendocrine tumors. Clinically, g-NETs are mainly classified into three types. Type I and type II are associated with chronic atrophic autoimmune gastritis[9] and gastrinoma-related Zollinger-Ellison syndrome (ZES) leading to hypergastrinemia, while type III is typically sporadic tumors associated with normal gastrin levels and poor prognosis. Although type 1 g-NETs caused by AAG are usually well-differentiated, studies have reported that 8%-23% of type 1 g-NETs extending into the deep submucosal layer may metastasize to regional lymph nodes or even to the liver. Furthermore, 3% of patients may develop neuroendocrine carcinoma, highlighting the need for appropriate attention.

Due to the destruction of gastric glands (including parietal and chief cells) in AAG patients, there is a deficiency in intrinsic factor, gastric acid, and a decrease in pepsinogen I (PG-I) levels. Insufficient gastric acid secretion leads to a compensatory increase in gastrin secretion by G cells in the gastric antrum, which acts on receptors present in enterochromaffin-like cells (ECL) in the gastric body and fundus, promoting ECL cell proliferation. Prolonged stimulation by hypergastrinemia can result in the development of ECL cell tumors, namely type 1 g-NETs. Considering the close association between type 1 g-NETs and AAG, primarily related to hypergastrinemia resulting from reduced gastric acid secretion, it is hypothesized that supplementation with gastric acid could provide negative feedback regulation of gastrin, reducing the risk of type 1 g-NET development in AAG patients. This study aims to investigate the impact of Betaine hydrochloride(BHCL) on gastrin levels in AAG patients, thus exploring a simple and cost-effective method to reduce the risk of type 1 g-NETs in AAG patients.

ELIGIBILITY:
Inclusion Criteria:

- 1) Patients diagnosed with autoimmune atrophic gastritis at the First Affiliated Hospital of Zhengzhou University, using the diagnostic criteria from the "Guidelines for the Diagnosis and Treatment of Chronic Gastritis in China (2022, Shanghai)" for the diagnosis of atrophic gastritis, combined with serum gastrin, PCA, or IFA for the diagnosis of autoimmune atrophic gastritis.

2) Patients who have signed the informed consent form for the clinical trial.

Exclusion Criteria:

* 1) Patients with Betaine hydrochloride allergies. 2) Patients with gastric ulcers, gastroesophageal reflux disease, or cholelithiasis, as the administration of acid agents may worsen the condition or cause discomfort.

  3) Patients with gastrinomas or other conditions that can cause elevated gastrin levels, apart from autoimmune atrophic gastritis.

  4) Patients who are unable to provide informed consent or sign the informed consent form.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
The difference in serum gastrin (1 month) | 1month
  Comparison of the difference in serum gastrin before and after the trial within each group.

SECONDARY OUTCOMES:
the adverse reaction rates | 3 months
  Adverse reaction rate = Number of patients with adverse reactions in each group / Number of patients examined in each group.
The difference in serum gastrin (3 month) | 3 months
  Comparison of the difference in serum gastrin before and after the trial within each

CONTACTS AND LOCATIONS:
Overall Officials: Jianning Yao, Dr., Study Chair — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

REFERENCES:
- [Background] Toh BH, Chan J, Kyaw T, Alderuccio F. Cutting edge issues in autoimmune gastritis. Clin Rev Allergy Immunol. 2012 Jun;42(3):269-78. doi: 10.1007/s12016-010-8218-y. PMID 21174235
- [Background] Anagnostopoulos GK, Ragunath K, Shonde A, Hawkey CJ, Yao K. Diagnosis of autoimmune gastritis by high resolution magnification endoscopy. World J Gastroenterol. 2006 Jul 28;12(28):4586-7. doi: 10.3748/wjg.v12.i28.4586. PMID 16874879
- [Background] Martinelli TM, van Driel IR, Alderuccio F, Gleeson PA, Toh BH. Analysis of mononuclear cell infiltrate and cytokine production in murine autoimmune gastritis. Gastroenterology. 1996 Jun;110(6):1791-802. doi: 10.1053/gast.1996.v110.pm8964405.
- [Background] Rustgi SD, Bijlani P, Shah SC. Autoimmune gastritis, with or without pernicious anemia: epidemiology, risk factors, and clinical management. Therap Adv Gastroenterol. 2021 Aug 31;14:17562848211038771. doi: 10.1177/17562848211038771. eCollection 2021. PMID 34484423
- [Background] Minalyan A, Benhammou JN, Artashesyan A, Lewis MS, Pisegna JR. Autoimmune atrophic gastritis: current perspectives. Clin Exp Gastroenterol. 2017 Feb 7;10:19-27. doi: 10.2147/CEG.S109123. eCollection 2017. PMID 28223833
- [Background] Lenti MV, Rugge M, Lahner E, Miceli E, Toh BH, Genta RM, De Block C, Hershko C, Di Sabatino A. Autoimmune gastritis. Nat Rev Dis Primers. 2020 Jul 9;6(1):56. doi: 10.1038/s41572-020-0187-8. PMID 32647173
- [Background] Niederle MB, Hackl M, Kaserer K, Niederle B. Gastroenteropancreatic neuroendocrine tumours: the current incidence and staging based on the WHO and European Neuroendocrine Tumour Society classification: an analysis based on prospectively collected parameters. Endocr Relat Cancer. 2010 Oct 5;17(4):909-18. doi: 10.1677/ERC-10-0152. Print 2010 Dec. PMID 20702725
- [Background] Delle Fave G, O'Toole D, Sundin A, Taal B, Ferolla P, Ramage JK, Ferone D, Ito T, Weber W, Zheng-Pei Z, De Herder WW, Pascher A, Ruszniewski P; Vienna Consensus Conference participants. ENETS Consensus Guidelines Update for Gastroduodenal Neuroendocrine Neoplasms. Neuroendocrinology. 2016;103(2):119-24. doi: 10.1159/000443168. Epub 2016 Jan 19. No abstract available. PMID 26784901
- [Background] Vannella L, Sbrozzi-Vanni A, Lahner E, Bordi C, Pilozzi E, Corleto VD, Osborn JF, Delle Fave G, Annibale B. Development of type I gastric carcinoid in patients with chronic atrophic gastritis. Aliment Pharmacol Ther. 2011 Jun;33(12):1361-9. doi: 10.1111/j.1365-2036.2011.04659.x. Epub 2011 Apr 15. PMID 21492197
- [Background] Borch K, Ahren B, Ahlman H, Falkmer S, Granerus G, Grimelius L. Gastric carcinoids: biologic behavior and prognosis after differentiated treatment in relation to type. Ann Surg. 2005 Jul;242(1):64-73. doi: 10.1097/01.sla.0000167862.52309.7d. PMID 15973103
- [Background] La Rosa S, Inzani F, Vanoli A, Klersy C, Dainese L, Rindi G, Capella C, Bordi C, Solcia E. Histologic characterization and improved prognostic evaluation of 209 gastric neuroendocrine neoplasms. Hum Pathol. 2011 Oct;42(10):1373-84. doi: 10.1016/j.humpath.2011.01.018. Epub 2011 May 4. PMID 21531442
- [Background] Qvigstad G, Falkmer S, Westre B, Waldum HL. Clinical and histopathological tumour progression in ECL cell carcinoids ("ECLomas"). APMIS. 1999 Dec;107(12):1085-92. doi: 10.1111/j.1699-0463.1999.tb01513.x. PMID 10660138
- [Background] Toh BH. Pathophysiology and laboratory diagnosis of pernicious anemia. Immunol Res. 2017 Feb;65(1):326-330. doi: 10.1007/s12026-016-8841-7. PMID 27538411
- [Background] Grozinsky-Glasberg S, Alexandraki KI, Angelousi A, Chatzellis E, Sougioultzis S, Kaltsas G. Gastric Carcinoids. Endocrinol Metab Clin North Am. 2018 Sep;47(3):645-660. doi: 10.1016/j.ecl.2018.04.013. Epub 2018 Jul 11. PMID 30098721
- [Background] Basuroy R, Srirajaskanthan R, Prachalias A, Quaglia A, Ramage JK. Review article: the investigation and management of gastric neuroendocrine tumours. Aliment Pharmacol Ther. 2014 May;39(10):1071-84. doi: 10.1111/apt.12698. Epub 2014 Mar 13. PMID 24628514

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-30): https://cdn.clinicaltrials.gov/large-docs/00/NCT06272500/Prot_SAP_002.pdf
  • Informed Consent Form (2024-01-30): https://cdn.clinicaltrials.gov/large-docs/00/NCT06272500/ICF_003.pdf